CLINICAL TRIAL: NCT06023849
Title: Trans Caesarean Intra Uterine Contraceptive Device Insertion Versus Conventional Postpartum 6 Weeks Insertion
Acronym: IUDinsertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed M.Osman, doctor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Trans CS IUCD insertion
Record Dates: First submitted 2023-08-06; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: IUD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPIUD (Active Comparator): trans cesarean IUD insertion immediately post placental
  Interventions: Device: IUD insertion
- interval (Active Comparator): IUD insertion 6 weeks interval post-partum
  Interventions: Device: IUD insertion

INTERVENTIONS:
Device: IUD insertion — Trans Caesarean Intra Uterine Contraceptive Device Insertion and Conventional Postpartum 6 Weeks Insertion

SUMMARY:
To compare immediate post-placental intrauterine contraceptive device insertion versus conventional placement at 6 weeks interval (often referred to as delayed or interval insertion) as regard to:-

1. Patient satisfaction.
2. Expulsion rate.
3. Complications

DETAILED DESCRIPTION:
Until the 1960s, Intrauterine devices (IUCDs) and condoms were the only artificial methods for the control of fertility. Nowadays ,despite the presence of 12 contraceptive methods which include 9 modern methods (pill, IUD, injectable, implant, vaginal methods (diaphragm and contraceptive foam or jelly), male condom, female sterilization, male sterilization, and emergency contraception) and 3 traditional methods (periodic abstinence, withdrawal, and prolonged breastfeeding , the insertion of an IUCD still the second most prevalent method of family planning used worldwide (13.6%), after female sterilization (20.5%), among women of reproductive age who are married or cohabiting.

In Egypt, Egypt Demographic and Health Survey 2014 findings revealed that 59 percent of currently married women in Egypt are currently using a contraceptive method. The most widely used method is the IUD, followed by the pill and injectables. Thirty percent of currently married women are using the IUD, 16 percent are relying on the pill, and 9 percent are employing injectables. Relatively small proportions of women are using other modern methods, e.g., 1 percent reported currently using female sterilization. Two percent of women report use of traditional methods.

There are two ways used in IUD insertion, in the postpartum period or immediate post-placental IUD insertion, in which the insertion of IUD occurs within ten minutes after placenta delivery and after the puerperium (after puerperal or interval period). Intrauterine device insertion during cesarean section was first introduced in 1967 by Zerzavy by suturing the IUD to the posterior uterine fundus. Research in China and Belgium introduced post-placental IUD insertion technique during cesarean delivery with placed an IUD as high as possible in the fundus without suturing the fundus wall.

Intrauterine device insertion during early postpartum period is the most effective reversible contraceptive methods for many mothers because the contraception motivation is high, and it doesn't interfere with breast feeding. On the other hand, without an effective contraception in the first six weeks, woman may be accidentally pregnant. Hence, the mother prefers to insert IUD during cesarean delivery.

As cesarean section (CS) rates are rising in all countries, IUD insertion at the time of CS creates an opportunity to increase access to long-acting reversible contraception methods. Conversely, a previous CS scar may deter access to interval insertion of an IUD if a previous CS may result in difficulty with insertion and/or future IUD problems.

Inserting an IUD at the time of CS is a very attractive option; It adds very little time and cost to the procedure. The patient does not have to come back especially for follow-up, and there is no risk of primary perforation (secondary perforation is possible) as it is performed under direct vision.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40years.
* Full term pregnancies delivered by cesarean section.
* Desire to have intrauterine contraceptive device (Cu T) as a contraceptive option.
* Agree to participate in the study.

Exclusion Criteria:

* Allergy to copper.
* Ante- or intra-partum hemorrhage.
* Ruptured of membranes for more than 18 h prior to delivery or Chorioamnionitis.
* Known uterine abnormalities e.g., Bicornuate/septate Uterus, uterine myoma.
* History of ectopic pregnancy.
* Desire for pregnancy within 1 year of delivery.
* Intrapartum fever >38 c.
* Sever thrombocytopenia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
1-Patient satisfaction and complication. | 6 months
  assessment of patient satisfaction using a questionnaire as follow:
  * Will you use the same method of contraception after the next delivery?
  * Will you recommend the same method to your fellows?
  * Are you happy or not with this procedure? give score from 1 to 10, 1 mean you are very unhappy while 10 mean you are very happy.
  * have you developed any complication?

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicin, Asyut, Egypt

REFERENCES:
- [Background] Hem E, Bordahl PE. Max Sanger - father of the modern caesarean section. Gynecol Obstet Invest. 2003;55(3):127-9. doi: 10.1159/000071524. PMID 12865589